CLINICAL TRIAL: NCT04961099
Title: Phase I Clinical Study on the Safety, Tolerance, Efficacy and Pharmacokinetics of Repeated Intratympanic HY01 in Patients With Sudden Sensorineural Hearing Loss
Brief Title: Phase I Clinical Study of HY01 in Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heyu (Suzhou) Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HY01-I-001
Record Dates: First submitted 2021-06-13; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Sudden Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sudden

STUDY DESIGN:
Intervention Model Description: HY01 will be administrated on D1, D4 and D7, and no other drugs or treatments will be given during the trial period (D1-30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose group (Experimental): low-dose group: HY01 10mg（20mg/ml）
  Interventions: Drug: HY01
- high-dose group (Experimental): high-dose group: HY01 20mg（40mg/ml）
  Interventions: Drug: HY01

INTERVENTIONS:
Drug: HY01 — low-dose group: HY01 10mg（20mg/ml）, administrated on D1, D4 and D7 high-dose group: HY01 20mg（40mg/ml）, administrated on D1, D4 and D7

SUMMARY:
Phase I clinical study on the safety, tolerance, efficacy and pharmacokinetics of repeated intratympanic HY01 in patients with sudden sensorineural hearing loss. In this study, low-dose group and high-dose group were designed, 6 cases in each group.

DETAILED DESCRIPTION:
The incidence rate of sudden deafness is increasing year by year, which can cause severe hearing loss. Intratympanic HY01 can increase the local drug concentration in the ear, which is equal to or better than that in the treatment of sudden sensorineural hearing loss, and reduce the systemic drug concentration at the same time. It has obvious clinical value for the treatment of hormone forbidden population.

HY01 is one of glucocorticoid drugs. In this study, we designed low-dose group and high-dose group of HY01, and enrolled 6 patients with sudden sensorineural hearing loss for salvage therapy in each group. HY01 will be administrated on D1, D4 and D7 . The trial will be ended 30 days after the first administration.

After determining the safety of low-dose, the patients in the high-dose group will be enrolled. The safety observation indexes included systemic Routine Indexes and otology indexes, and the efficacy and pharmacokinetics were observed at the same time.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese subjects were 18-65 years old (including boundary value), male and female were not limited;
2. Patients with unilateral sudden deafness;
3. At least 7 days after the last medication (according to the guidelines for diagnosis and treatment of sudden deafness, the drugs allowed to be used include glucocorticoids, batroxobin, neurotrophic drugs (such as Mecobalamin, neurotrophic factors, etc.), antioxidants (such as lipoic acid, Ginkgo biloba extract, etc.) and lidocaine) ;
4. The hearing recovery of patients with sudden deafness after initial treatment is less than 15dB or less than 50% of the hearing of the affected ear or the healthy ear before the onset of the disease ;
5. 19≤BMI<26kg/m2；
6. After at least one course of standard treatment (according to the guidelines for diagnosis and treatment of sudden deafness, systemic hormone combined with other drugs) ;
7. The informed consent was signed before the trial, and the trial content, process and possible adverse reactions were fully understood.

Exclusion Criteria:

- Ear diseases

1. Patients with bilateral sudden deafness;
2. The initial treatment was intratympanic glucocorticoid;
3. The average hearing threshold of healthy ear was more than 25 dB;
4. Patients with previous or current ear related diseases may affect the judgment of adverse events, including but not limited to chronic ear infection, cholesteatoma, Meniere's disease, otosclerosis, fluctuating hearing loss, acoustic trauma, autoimmune hearing loss, radiation-induced hearing loss, syphilitic deafness, endolymphatic hydrops, hearing loss caused by otological surgery Suspected retrocochlear lesions, suspected perilymph fistula or membrane rupture, perilymph fistula or barotrauma, acoustic neuroma, synchronous tinnitus (possibly caused by glomus jugulare tumor), skull, face or temporal bone abnormalities;
5. Subjects with congenital deafness and hereditary deafness;
6. Treatment history of ototoxicity drugs within 6 months, such as chemotherapy, loop diuretics, aminoglycosides, quinine, high-dose aspirin, etc;
7. Subjects considered unsuitable for this clinical study.

   Systemic diseases
8. Previous or current contraindications to glucocorticoids include hypertension, thrombosis, myocardial infarction, gastric and duodenal ulcer, visceral surgery, psychosis, electrolyte metabolism abnormality, glaucoma;
9. Previous or current patients with glucocorticoid caution include infection, ulcerative colitis, diverticulitis, postoperative enterostomy, liver cirrhosis, renal dysfunction, epilepsy, migraine, myasthenia gravis, osteoporosis, hypothyroidism, ocular herpes simplex, chickenpox or measles, recent live attenuated vaccine, latent tuberculosis or old tuberculosis Hepatitis B virus carriers;
10. Corticosteroid related psychiatric reactions;
11. It is forbidden to use this product for allergic patients, and it should be used with caution for subjects with allergic history to adrenocortical hormone drugs;
12. Subjects with positive TB history or tuberculin test (PPD);
13. Type 1 and type 2 diabetes;
14. pancreatitis;
15. Suffering from rheumatic diseases, such as rheumatoid arthritis, scleroderma, lupus, etc;
16. Previous or current use of chemotherapy or immunosuppressive drugs;
17. Active herpes zoster;
18. Those who had taken any medicine other than sudden deafness within 14 days before the first administration;
19. There was a history of alcohol abuse and drug abuse in one year before screening;
20. Those who had participated in any clinical trial within 3 months before the first administration of the trial;
21. Blood donation or blood loss ≥ 200ml within 3 months before the first administration;
22. Those who do not agree to avoid using alcohol, tobacco or caffeinated drinks within 24 hours before and during the trial, or to avoid strenuous exercise, or to avoid other factors affecting drug absorption, distribution, metabolism and excretion;
23. Pregnant or lactating women, or those whose plasma hCG test was positive, or those who could not or did not take contraceptive measures approved by the researcher within 6 months from the study period to the end of the study according to the guidance of the researcher;
24. Serological tests or other tests showed that subjects with positive hepatitis B, HCV, syphilis and AIDS were positive.
25. Subjects considered unsuitable for this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of HY01 | Throughout the study approximately 30 days
  AEs and SAEs

SECONDARY OUTCOMES:
Hearing improvement | Day 30
  Change from baseline to Day 30 of Pure Tone Audiometry(250 Hz、500 Hz、1000 Hz、2000 Hz、3000 Hz、4000 Hz、8000 Hz)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Pin, Doctor, Study Director — Shanghai Central Hospital
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No